CLINICAL TRIAL: NCT01525004
Title: Randomized, Double Blind, Comparison of Standard Dose Trivalent Inactivated Influenza Vaccine in Pediatric Solid Organ Transplant Patients
Brief Title: Standard Dose Versus High-Dose Inactivated Flu Vaccine in Pediatric Solid Organ Transplant Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of Pittsburgh (Other); MCM Vaccines B.V. (Industry)
Responsible Party: Principal Investigator, Natasha Halasa, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 111069 - IRB
Record Dates: First submitted 2011-10-14; First posted 2012-02-02 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Pediatric Solid Organ Transplant Patients
Keywords: Solid organ transplant; Flu vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard dose trivalent inactivated influenza vaccine (Active Comparator)
  Interventions: Drug: Standard dose trivalent inactivated influenza vaccine
- High-Dose trivalent inactivated influenza vaccine (Experimental)
  Interventions: Drug: High-Dose trivalent inactivated influenza vaccine

INTERVENTIONS:
Drug: High-Dose trivalent inactivated influenza vaccine — 0.5 mL of high-dose trivalent inactivated influenza vaccine, either one dose or 2 based on whether the patient has previously received standard dose trivalent inactivated influenza vaccine.
  Arms: High-Dose trivalent inactivated influenza vaccine
Drug: Standard dose trivalent inactivated influenza vaccine — 0.5 mL standard dose trivalent inactivated influenza vaccine, either one dose or 2 based on whether the patient has previously received standard dose trivalent inactivated influenza vaccine
  Arms: Standard dose trivalent inactivated influenza vaccine

SUMMARY:
This is a phase I trial in which the both the safety and immunogenicity of the standard dose flu vaccine will be compared with high dose flu vaccine in children that have undergone solid organ transplantation (SOT).

DETAILED DESCRIPTION:
A prospective, randomized, double-blind phase 1 safety and immunogenicity study of the HD compared with the SD TIV in pediatric patients between the ages of three and 17 yr that have undergone SOT (Clin-Trials.gov. NCT01525004) was conducted. Subjects were randomized in a 2:1 fashion to receive 0.5 mL of either the HD (60 μg) or SD (15 μg) TIV intramuscularly. Subjects <9 yr of age received either one or two doses of the vaccine based on ACIP recommendations [19]. The study was approved by Institutional Review Boards at both institutions (Vanderbilt University, Nashville, TN, and the University of Pittsburgh, Pittsburgh, PA) and conducted during the 2011-2012 influenza season. Subjects were randomly allocated to either the HD or SD group by a computer-generated allocation system. Participants, their families, and research staff who performed clinical evaluations remained blinded to the child's assigned dosage, while designated unblinded nurses administered the requisite vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric SOT patients (kidney, liver, heart, lungs, intestine, and/or multi-visceral)
* Must be at least 6 months after transplant.
* 3-17 years of age, inclusive.
* Available for duration of study.
* Parent or guardian able to be reached by phone.

Exclusion Criteria:

* History of hypersensitivity to previous influenza vaccination or severe hypersensitivity to eggs/egg protein.
* History of Guillian-Barre syndrome.
* Receipt of rituximab within the past one year.
* Rejection treatment with intravenous steroid bolus within 30 days.
* Rejection treatment with monoclonal antibody or antilymphocyte preparation (e.g. Alemtuzumab, Muromonab-CD3, etc.) within 90 days.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Have any condition that the investigator believes may interfere with successful completion of the study.
* History of received 2011-2012 influenza vaccine.
* Pregnant female.
* History of proven influenza disease after September 1, 2011.
* History of known infection with HIV, hepatitis B, or hepatitis C.
* History of known latex hypersensitivity.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety profile of high dose trivalent inactivated influenza vaccine to standard dose trivalent inactivated influenza vaccine in pediatric solid organ transplant patients | 6-9 months
  We will record local and systemic reactions after each vaccination for seven days. Patients will fill out a diary card. We will collect adverse events for 28 days and SAE for 6 months.

SECONDARY OUTCOMES:
Humoral immune responses of pediatric Solid Organ Transplant patients to influenza virus antigens included in trivalent inactivated influenza vaccine after high and standard doses of trivalent inactivated influenza vaccine. | 12 months
  We will measure HAI titers. We will calculate the perecet of subjects who acheive HAI titers greater than and equal to 1:40 and those with 4-fold increase. We will also calculate GMTs.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Halasa, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt University, Nashville, Tennessee, United States